CLINICAL TRIAL: NCT03026205
Title: Evaluation of the Safety, Tolerability and Pharmacokinetics of Single and Multiple Doses of Orally Administered ARMS-I Administered in Healthy Adults, Aged 18-45 Years
Brief Title: ARMS-I (a Formulation of Cetylpyridinium Chloride -CPC)
Acronym: ARMS-I
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Collaborators: ProMedica Health System (Other); The University of Toledo (Unknown); ARMS Pharmaceutical LLC (Unknown); Pediatric Pharmacology Research Center (Unknown)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-191
Record Dates: First submitted 2017-01-12; First posted 2017-01-20 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Viral Upper Respiratory Tract Infection
MeSH Terms: interventions — Cetylpyridinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): ARMS-I dosage of 0.75 mg will be sprayed orally in the mouth once as a single dose of four sprays on Day 1, and then three times a day starting on Day 3 for 4 Days.
  Interventions: Drug: ARMS-I

INTERVENTIONS:
Drug: ARMS-I
  Other Names: Cetylpyridinium Chloride

SUMMARY:
This is a single center study to evaluate the pharmacokinetics of ARMS-I a formulation that incorporates cetylpyridinium chloride (CPC), administered once as a single dose of three sprays orally, followed by multiple dosing (3x daily oral sprays) over days 3-6 and then a repeat pharmacokinetic study during the final oral dose administered as the first dose on day 7 to ascertain CPC accumulation.

DETAILED DESCRIPTION:
ARMS Pharmaceuticals LLC intends to apply for approval of ARMS-I as a prescription drug for the prevention of influenza, rhinovirus and RSV (collectively, "vURTI's). The company plans on confirming the limited systemic bioavailability, through conducting a study to characterize the pharmacokinetics of ARMS-I administered orally in healthy adults. The primary objective of the study is to determine the pharmacokinetics of ARMS-I following oral administration to healthy subjects. Specifically, investigators will assess whether there is measurable systemic exposure and if so, to determine the plasma and pharyngeal fluid pharmacokinetic characteristics of ARMS-I after single and multiple oral dosing. The secondary objective will be to evaluate the safety and tolerability of ARMS-I.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 45 years of age, inclusive
* Ability to understand the consent process and procedures
* Informed consent obtained and signed
* Comprehension of the protocol, which will be determined by the recruiter after explaining the procedures
* Subjects agree to be available for all study visits. Subjects will be asked if they have any travel plans, and whether staff could use alternate contact information that will be provided.
* General good health as determined by the Study Physician, without current medical illness or clinically significant abnormal physical examination findings that classify the subject as other than healthy
* Negative urine pregnancy test at screening and a negative urine pregnancy test on the day of initial pharmacokinetic sampling for all female subjects of child bearing potential
* Negative urine toxicity screen for marijuana, cocaine metabolites, amphetamines, opiates, PCP, barbiturates, benzodiazepines
* Negative breathalyzer for alcohol
* Body mass index (BMI) between 18 and 35 (inclusive) [weight (kg)]/ [height (m)2]
* No tobacco/nicotine use for at least 3 months prior to study enrollment
* No oral disease or lesions
* Agreement to refrain from eating or drinking except for water for 8 hours prior to drug administration and eating or drinking anything for 4 hours after dosing on the days of pharmacokinetic sampling
* Agreement by subjects with reproductive potential to use an adequate method of contraception during the study and for one week after study drug administration. Female subjects must agree to the use of TWO reliable methods of contraception while receiving study drug and for 4 weeks after study drug administration, which can include: condoms, spermicidal gel, diaphragm, hormonal or non-hormonal intrauterine device, surgical sterilization, oral contraceptive pill, depot progesterone injections, and sexual abstinence. If a male subject is sexually active, the subject and his partner must agree to use at least one of the above listed contraceptive methods.
* If the subject uses abstinence and becomes sexually active during the study, they must agree to use TWO forms of contraception if female and ONE if male, of the above listed contraceptive methods.

Exclusion Criteria:

* Hypertension with confirmed systolic blood pressure >140 mmHg or confirmed diastolic blood pressure >90 mmHg, measured after 10 - 15 minutes of rest
* Morbid obesity (BMI>35)
* Current diagnosis of pulmonary disease including asthma or COPD, which has required use of asthma medications within the past year
* History of or current diagnosis of diabetes
* Autoimmune disorder, such as systemic lupus erythematosus, Wegener's disease, or rheumatoid arthritis, among other conditions
* History of malignancy except low-grade skin cancer, (i.e., basal cell carcinoma which has been surgically cured)
* Chronic renal, hepatic, or pulmonary disease condition that could interfere with the absorption of the study drug (e.g., surgical resection of significant proportions of the stomach or bowel, gastric bypass, gastric banding, irritable bowel syndrome, inflammatory bowel disease)
* Blood donation within the previous 6 weeks
* History of cardiac rhythm abnormality
* History of prolonged QT interval
* Prolongation of QTcB interval (i.e., confirmed QTcB interval >450 milliseconds)
* Clinically significant abnormal electrocardiogram at screening in the judgment of the investigator, or based on the formal ECG reading; history of any cardiac abnormalities, including conduction abnormalities such as Wolff-Parkinson-White Syndrome, dysrhythmias, or coronary artery disease
* Laboratory values outside the normal ranges in Appendix for the following tests: blood cell counts (white blood cell counts [WBC], hemoglobin, platelets), serum chemistry (sodium, potassium, calcium, chloride, CO2, creatinine, glucose, BUN, AST, AP, ALT, total bilirubin, protein, albumin, amylase), urinalysis for glucose, protein and blood (with proviso for re-testing menstruating females). If CK is above normal range at baseline, but not clinically significant, the subject can be included.
* Positive serology results for HIV, HBsAg, or HCV infections
* Febrile illness with temperature documented >38°C within 7 days of dosing
* Pregnancy or breastfeeding
* Known allergic reactions to study drug components, including ingredients present in the formulation.
* Treatment with another investigational drug within 30 days of dosing
* Lack of ability to fully understand the informed consent form. This will be determined by the recruiter/interviewer after explaining the consent and observing the subject reading the consent.
* Ingestion of prescription medications, grapefruit juice, or St John's Wort starting 14 days or 5 half-lives before dosing, whichever is longer. Women may use oral contraceptives.
* Ingestion of herbal supplements or over-the-counter medications starting 7 days before dosing
* Use of any form of tobacco, including cigarette smoking, pipe smoking, or oral tobacco; if a former smoker or tobacco user, the subject must not have used tobacco for 90 days before screening
* Any specific condition that, in the judgment of the Principal Investigator, precludes participation because it could affect subject safety
* History of current use of narcotics, or recreational drug use.
* Use of > 7 alcoholic beverages within 1 week
* Use of any other intra-oral product (especially antiseptic) except for dental hygiene
* Use of any systemic antimicrobial agent within 30 days of screening
* Prior or current history of seasonal allergies, chronic sinusitis or rhinitis
* Presence of oral lesions
* Use of dentures
* Dental treatment currently in progress (implants, root canals, complex restorative procedures)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Plasma and pharyngeal fluid concentrations | 1 week
  Plasma and pharyngeal fluid concentrations of the active ingredient of ARMS-I (CPC) will be measured before and at multiple time points after the oral administration. If plasma concentrations are measureable (above the LLOQ) then the assessed PK parameters will include Cmax
Plasma and pharyngeal fluid concentrations | 1 week
  If plasma concentrations are measureable (above the LLOQ) then the assessed PK parameters will include AUC0-t
Plasma and pharyngeal fluid concentrations | 1 week
  If plasma concentrations are measureable (above the LLOQ) then the assessed PK parameters will include AUC0-24
Plasma and pharyngeal fluid concentrations | 1 week
  If plasma concentrations are measureable (above the LLOQ) then the assessed PK parameters will include C24
Plasma and pharyngeal fluid concentrations | 1 week
  If plasma concentrations are measureable (above the LLOQ) then the assessed PK parameters will include C48
Plasma and pharyngeal fluid concentrations | 1 week
  If plasma concentrations are measureable (above the LLOQ) then the assessed PK parameters will include Cl/F
Plasma and pharyngeal fluid concentrations | 1 week
  If plasma concentrations are measureable (above the LLOQ) then the assessed PK parameters will include Tmax
Plasma and pharyngeal fluid concentrations | 1 week
  If plasma concentrations are measureable (above the LLOQ) then the assessed PK parameters will include t½

SECONDARY OUTCOMES:
Frequency of adverse events | 30 days from point of enrollment
  The frequency of adverse events (both solicited and unsolicited) will be assessed on a continuous basis throughout the study via safety assessments, observation direct participant reporting, and specific adverse reaction inquiry. Physical examinations, vital signs, ECG's, hematology, serum chemistries, coagulation studies and urinalysis will also be used to assess safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Blumer, PhD, MD, Principal Investigator — Professor, University of Toledo
Locations (1):
- ProMedica Health System, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No